CLINICAL TRIAL: NCT06338020
Title: Effects of Adaptive Variable-resistance Training on Chemotherapy-induced Sarcopenia, Fatigue, and Functional Restriction in Pediatric Survivors of Acute Lymphoblastic Leukemia: A Large-scale Randomized Controlled Trial
Brief Title: Adaptive Variable-Resistance Training in Pediatric Survivors of Acute Lymphoblastic Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ragab Kamal Elnaggar, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/0022/0042
Record Dates: First submitted 2024-03-23; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: A prospective, dual-arm, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: This was a single-blind protocol. The researcher who collected the data was blind to the allocation of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adaptive-VRT (Experimental): Participants in this group received the adaptive variable-resistance training program in besides the standard physical therapy care.
  Interventions: Other: Adaptive variable-resistance training
- Standard Physical Therapy (Active Comparator): Participants in this group received the standard exercise program.
  Interventions: Other: Standard physical therapy

INTERVENTIONS:
Other: Adaptive variable-resistance training — The training was conducted thrice weekly for eight successive weeks under the close supervision of a licensed pediatric physical therapist in accordance with the safety performance guidelines defined by the American Academy of Pediatrics and the US National Strength and Conditioning Association.
  The training protocol included maximum voluntary concentric knee flexor/extensor actions. Three sets of five to 10 repetitions of maximum-effort concentric action at angular speeds of 240, 180, and 120 degrees/second.
  The training started with a 10-minute warm-up exercise and ended up with a 5-minute cool-down exercise.
  Arms: Adaptive-VRT
Other: Standard physical therapy — The program encompassed the standard exercises for survivors of ALL (flexibility, graduated active strengthening, and conditioning exercises). The training was conducted for 45 minutes, two times a week for six successive weeks.
  Arms: Standard Physical Therapy

SUMMARY:
This study was designed to investigate the effect of eight weeks of adaptive variable-resistance training (Adaptive-VRT) on chemotherapy-induced sarcopenia, fatigue, and functional restrictions in a convenience sample of pediatric survivors of acute lymphoblastic leukemia (ALL). Sixty-two pediatric survivors of ALL were randomly allocated to the experimental group (n = 31, received the adaptive variable-resistance training) or the Control group (n = 31, received standard physical therapy care). Both groups were assessed for muscle mass, strength, fatigue, and functional capacity before and after treatment.

DETAILED DESCRIPTION:
Sixty-two pediatric survivors of ALL participated in the study. They were recruited from the Pediatric Oncology/Hematology departments of three referral hospitals in Riyadh region, Saudi Arabia. They were between 12 and 18 years old, completed chemotherapy, had secondary sarcopenia, had normal cardiac structure and function, had no lower limb deformities, and did not engage in regular exercise regimens. They were excluded if they had secondary cancers, neurodegenerative impairments affecting memory, attention, or executive functioning, or neuro-musculoskeletal conditions likely to impede the training like recurrent intensive cramps or impaired proprioceptive functions.

Outcome measures

1. Muscle thickness: the thigh muscle thickness was assessed using a standard high-resolution ultrasound imaging system.
2. Muscle strength: The peak concentric torque of the right and left quadriceps was measured through an isokinetic dynamometer.
3. Fatigue: the general fatigue perception was evaluated using the Pediatric Quality of Life Inventory-Multidimensional Fatigue Scale.
4. Functional capacity: Three tests were used; the 6-minute walk test, the timed up and down stairs test, and the 4x10 meter Shuttle Run test.

The experimental group received an adaptive-VRT program, three times a week, for six consecutive weeks, in conformity with the National Strength and Conditioning Association guidelines and American Academy of Pediatrics safety standards. The training protocol included maximum voluntary concentric knee flexor/extensor actions through a motion range between 10 and 90 degrees. Three sets of five to 10 repetitions at angular speeds of 240, 180, and 120 degrees/second were performed. The training started with a warm-up for 10 minutes and ended with a cool-down for 5 minutes.

The control group received the standard exercise program, 45 minutes per session, three times a week, for eight consecutive weeks. The program consisted of flexibility exercise, manual/mechanical strength training, and moderate-intensity aerobic exercises on a treadmill or bicycle ergometer.

ELIGIBILITY:
Inclusion Criteria:

* Age between 12 and 18 years old
* Complete maintenance chemotherapy
* Secondary sarcopenia
* Normal cardiac structure and function
* Absence of lower limb deformities
* Not engaging in regular exercise regimens

Exclusion Criteria:

* Secondary cancers
* Neurodegenerative impairments affecting memory, attention, or executive functioning
* Neuro-musculoskeletal conditions are likely to impede the training.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Thigh muscle thickness | 2 months
  The distance between the anterior fascia of the rectus femoris muscle and the posterior fascia of the vastus intermedius muscle. It was measured using a high-resolution ultrasound imaging system.
Muscle strength | 2 months
  Muscle strength was indicated by the peak concentric torque of the knee extensors (Nm). It was measured using an Isokinetic Dynamometer.

SECONDARY OUTCOMES:
Fatigue | 2 months
  The general, sleep/rest, and cognitive fatigue perception was collectively measured using the Pediatric Quality of Life Inventory-Multidimensional Fatigue Scale. It is an 18-item scale measure fatigue in three domains (i.e., general, sleep/rest, and cognitive fatigue). Items are rated on a 5-point scale (0-4; where 0 means "never" and 4 means "almost always"). The total score was calculated and was then linearly transformed on a 0-100 scale. Higher scores indicate less fatigue and better functioning.
Six-minute walk test | 2 months
  This test identified the maximum distance (m) that each patient was able to cover over six minutes on a straight flat 30-m walkway, without running or jogging. Walking is regarded as more efficient in line with a longer distance coverage.
4x10 meter Shuttle Run test | 2 months
  This test measured the time (seconds) that each patient took to run forth and back a 10-meter track. Better performance is indicated by a shorter time.
Timed up and down stairs test | 2 months
  This test measured the time (seconds) that each patient took to climb up and down a 14-step stair flight (each 20 cm in height). Better performance is indicated by a shorter time.

CONTACTS AND LOCATIONS:
Overall Officials: Ragab K. Elnaggar, PhD, Principal Investigator — Prince Sattam Bin Abdulaziz University
Locations (1):
- Ragab K. Elnaggar, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elnaggar RK, Mahmoud WS, Abdrabo MS, Elfakharany MS. Effect of adaptive variable-resistance training on chemotherapy-induced sarcopenia, fatigue, and functional restriction in pediatric survivors of acute lymphoblastic leukemia: a prospective randomized controlled trial. Support Care Cancer. 2025 Feb 22;33(3):214. doi: 10.1007/s00520-025-09250-x. PMID 39985582